CLINICAL TRIAL: NCT03909880
Title: Effects of Kinesio Taping on Hand Proprioception, Reaction Time, Force Control and Corticomuscular Functional Connectivity
Brief Title: Kinesio Taping and Hand Sensorimotor Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YM108058E
Record Dates: First submitted 2019-02-11; First posted 2019-04-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2019-07

CONDITIONS: Healthy Adults
Keywords: kinesio taping, sensorimotor control
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Without Kinesio tape on the forearm
- Kinesio taping with neutral tension (Placebo Comparator): Kinesio tape with neutral tension on the forearm
  Interventions: Other: Kinesio tape
- Kinesio taping with additional 20% tension (Experimental): Kinesio tape with 20% additional tension on the forearm
  Interventions: Other: Kinesio tape

INTERVENTIONS:
Other: Kinesio tape — Kinesio tape (kinesio taping; kinesio holding corporation,USA) was placed on the skin above muscle belly of finger flexor. There were three types of taping:
  "Taping20 condition" - tape was pulled from the wrist to the proximal forearm. The two ends of the tape (~5 cm) were held by the therapist and the middle area was pulled 20% additional tension.
  "TapingN condition" - tape was pulled with neutral tension. "Control condition" - no taping.
  Arms: Kinesio taping with additional 20% tension; Kinesio taping with neutral tension

SUMMARY:
We explored the effect of Kinesio taping with different tension on hand force control, joint proprioception, reaction time and brain activity.

Healthy participants randomly received three wrist/finger flexor taping conditions: (1) taping with 20% additional tension (taping20), (2) taping with neutral tension (tapingN), and (3) without taping (control). Grip force, wrist joint angle, electroencephalogram and electromyogram were recorded during proprioception and force control tasks to determine the effects of Kinesio taping on sensorimotor control.

DETAILED DESCRIPTION:
Sensorimotor control involves the integration of sensory information in the brain to ensure appropriate joint position, force control and timing during movement. Kinesio taping can provide additional sensory input and improve sensorimotor control performance. Hand function is important in daily activities and fine control of the fingers and wrist is required in many sports. Therefore, we explore the effect of Kinesio taping with different tension on hand force control, joint proprioception, reaction time and brain activity.

This is an observational study with single-group repeated-measures design. Participants will be randomly received three wrist/finger flexor taping conditions: (1) taping with 20% additional tension (taping20), (2) taping with neutral tension (tapingN), and (3) without taping (control). Grip force, wrist joint angle, electroencephalogram and electromyogram were recorded during proprioception and force control tasks.Repeated-measures one-way analysis of variance and the Bonferroni post hoc comparison test determined the differences among the taping conditions. The Pearson correlation test determined the correlation between changes in motor performance and brain activities. Statistical significance was set at .05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults who are 20-40 years old

Exclusion Criteria:

1. Have irreversible injury on forearm, wrist or hand
2. Feel pain or any uncomfortable symptom on forearm, wrist or hand
3. Muscular disease on upper extremity in 6 months
4. Impaired sensation
5. Allergy to Kinesio tape
6. Neurological disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Joint position sense | measured immediately after the tape is applied
  The ability to accurately generate joint wrist flexion at 15 degree
Force sense | measured immediately after the tape is applied
  The ability to accurately generate 20% of maximal voluntary grip force
Reaction time | measured immediately after the tape is applied
  The ability to generate grip force as soon as hearing a beep sound
Corticomuscular coherence | measured immediately after the tape is applied
  Level of EEG and EMG synchronization in frequency domain when participants maintain 20% maximal voluntary contraction for 30 seconds, as an indicator of functional connectivity between motor cortex and muscle
EEG | measured immediately after the tape is applied
  Level of the power of EEG when participants maintain 20% maximal voluntary contraction for 30 seconds, as an indicator of synchronization/desynchronization of the motor cortex

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, Ph.D., Principal Investigator — Department of Physical Therapy and Assistive and Technology ,National Yang-Ming University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No